CLINICAL TRIAL: NCT03616444
Title: Clinical Evidence-based Evaluation of the Efficacy of Shenbai Granules in Preventing Recurrent Colorectal Adenomas After Polypectomy and Its Therapeutic Mechanism
Brief Title: A Randomized Clinical Trial of Shenbai Granules in Reducing Recurrence of Colorectal Adenoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Collaborators: Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Shanghai University of Traditional Chinese Medicine (Other); ShuGuang Hospital (Other); The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other); Changhai Hospital (Other); Beijing Friendship Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017YFC1700602
Record Dates: First submitted 2018-07-26; First posted 2018-08-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Gastroenterology
Keywords: colorectal adenoma; Clinical curative effect; Complementary and alternative medicine

STUDY DESIGN:
Intervention Model Description: colorectal adenomatous polyp patients after colonoscopy under colonoscopy
Who Masked: Participant, Investigator
Masking Description: A double-blind design is used in this study for the investigators and subjects. The blinding codes are separately sealed and stored by the independent third-party organization. Trial granules are randomly coded as subject unique identification codes, and used by each clinical site according to the assigned drug numbers and in the order of case enrollment. Clinical monitors and investigators must be blinded at all times.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM-Shenbai Granules (Experimental): Shenbai Granules: Hedyotis diffusa 10g, Sophorae flavescentis radix 4.5g, Codonopsis radix 7.5g, Atractylodis macrocephalae rhizoma 6g, Mume fructus 4.5g, Coptidis rhizoma 1.5g, Zingiberis rhizome praeparatum 3g, Coicis semen 10g.
  Orally, 1 sachet once, diluted in 150-200 ml of boiling water, 2 times a day.
  Interventions: Drug: Shenbai Granules
- TCM-Placebo (Placebo Comparator): It contains 5% SBG content, and the remaining ingredients are flavoring agents, starch and coloring agents. It is the same with SBG in appearance, smell and dosage form.
  Orally, 1 sachet once, diluted in 150-200 ml of boiling water, 2 times a day.
  Interventions: Drug: Shenbai Granules

INTERVENTIONS:
Drug: Shenbai Granules — In the first year, the trial granules will be started after enrollment for 3 months; In the second year, the trial granules will be started in the first 3 months; Each participant should have completed 6 months of trial granules.
  Other Names: placebo

SUMMARY:
This study evaluates Shenbai Granules in Prevention of Colorectal Adenomatous Polyp Recurrence After Colonoscopy.Half of participants will receive Shenbai Granules,while the other half will receive a placebo.

DETAILED DESCRIPTION:
There is no internationally recognized standard treatment for the prevention of recurrence of colorectal adenomatous polyps.

Based on TCM,previous studies have found that Shenbai Granules can significantly reduce the recurrence and deterioration rate of colorectal adenomatous polyps,reduce the proliferation of tumor cells and promote apoptosis of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. meet the colorectal adenomatous polyp diagnosis.
2. polypectomy under colonoscopy;Including snare polypectomy,endoscopic mucosal resection,endoscopic submucosal dissection.
3. aged 18-70.
4. sign informed consent.

Exclusion Criteria:

1. colonoscopy was reported, but no pathological findings were found.
2. patients with hereditary polyposis.
3. there is reliable evidence that the tumor has infiltrated into the intrinsic mucosal layer,or deep infiltration under the mucosa is suspected.
4. combined with colorectal malignancy or previous history of colorectal malignancy.
5. colonoscopy highly suggests inflammatory bowel disease.
6. pregnant and lactating women.
7. women who recently have a planning pregnant programme.
8. prone to bleeding and using anticoagulants.
9. patients with severe cardiovascular,pulmonary and cerebrovascular diseases and liver and kidney dysfunction (ALT and AST are two times higher than the upper limit of normal value in the laboratory of the center;Serum creatinine and urea nitrogen are 1.5 times higher than the upper limit of the normal value in the laboratory of the center.
10. unstable vital signs.
11. suspect or have a history of alcohol or drug abuse.
12. frequent changes in the working environment or other circumstances are likely to cause loss of interview.
13. drugs (aspirin, folic acid, vitamin D, calcium) with potential to treat colorectal adenomas have been used.
14. those who are participating in other clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 2 years
  The ratio of the number of patients with new adenoma detected by colonoscopy to the total number of cases in this group during follow-up.

SECONDARY OUTCOMES:
The detection rate of any polypoid lesions | 2 years
  The ratio of the number of patients with any polypoid lesions detected by colonoscopy to the total number of cases in this group during follow-up.
The detection rate of high-risk adenomas | 2 years
  The ratio of the number of patients with high-risk adenomas detected by colonoscopy to the total number of cases in this group during follow-up.
The detection rate of sessile serrated lesions | 2 years
  The ratio of the number of patients with sessile serrated lesions detected by colonoscopy to the total number of cases in this group during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yugen, PhD, Study Chair — Key members of the study
Locations (1):
- Affiliated Hospital of Nanjing University of TCM, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are restricted in availability due to patient confidentiality reasons.

REFERENCES:
- [Derived] Zhou Q, Chen YG, Xiao J, Chen TT, Liu JR, Zhou W, Li WZ, Wang Y, Zhang BP, Lin J, Meng FD, Gong B, Zheng GY, Han ST, Cheng HB. Traditional Chinese medicine (Xiaoai Jiedu Decoction) as an adjuvant treatment for prevention new colorectal adenomatous polyp occurrence in post-polypectomy: Study protocol for a randomized controlled trial. Medicine (Baltimore). 2019 Aug;98(31):e16680. doi: 10.1097/MD.0000000000016680. PMID 31374049

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT03616444/Prot_SAP_000.pdf